CLINICAL TRIAL: NCT02044510
Title: A Double Blind, Randomized Placebo Controlled Trial Evaluating the Urodynamic and Clinical Efficacy of Mirabegron Among Neurogenic Bladder Patients
Brief Title: Urodynamic and Clinical Efficacy of Mirabegron for Neurogenic Bladder Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow recruitment and small observed effect size
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Blayne Welk, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG193
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Urinary Bladder, Neurogenic
Keywords: Multiple Sclerosis; Spinal Cord Injuries; mirabegron; Urodynamics
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Multiple Sclerosis; Spinal Cord Injuries | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirabegron (Experimental): Patients randomised to this arm start with mirabegron 25mg PO daily for two weeks, and then at 2 weeks titrate to 50mg PO daily, and maintain that dose for the duration of the study (8 additional weeks).
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator): Inert placebo pill, matching active treatment pill.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron — Mirabegron 25mg PO daily for 2 weeks, with dose increase to Mirabegron 50mg PO daily for the remaining 8 weeks.
  Other Names: MYRBETRIQ
  Arms: Mirabegron
Drug: Placebo — Matched placebo capsules to the intervention arm
  Arms: Placebo

SUMMARY:
The proposed study is a randomized, double blind placebo controlled multicenter study to determine the effectiveness of mirabegron in the treatment of neurogenic bladder dysfunction. Patients will be randomized into one of two trial arms: mirabegron 25mg for two weeks, with escalation to 50mg for the remaining 8 weeks, or matched placebo capsule for two weeks, with placebo escalation for the remaining 8 weeks. Each of these trial arms will be stratified based on whether the patient is already taking an anticholinergic medication or not. The study will treat a total of 144 patients (72 with placebo, 72 with mirabegron). The study hypothesis is that mirabegron will result in a statistically superior (increased) urodynamic bladder capacity.

The study duration is 12 weeks, with a 1-4 week run in period where no active or placebo treatment will be administered. The primary outcome measure will be based on an increase in urodynamic bladder capacity. Secondary outcome measures will be additional urodynamic parameters, urinary symptom scales, urinary quality of life indices, and voiding diary results.

Patients who are over 18 years of age with a diagnosis of multiple sclerosis (MS) or spinal cord injury (SCI) will be eligible to participate. All eligible patients will have urodynamic studies performed within 4 weeks of trial enrollment, and at the end of study (week 9-10). Adverse events and study outcomes will be assessed at predefined study time points.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of traumatic or nontraumatic suprasacral spinal cord injury (SCI) or multiple sclerosis (MS, based on a neurologist assessment and/or the McDonald criteria)(28)
* Age >18 years
* Stable method of bladder management for >3months (either spontaneous or provoked voiding, or intermittent catheterization).
* Bothersome urinary symptoms (urinary frequency, urgency, or urgency incontinence based on standard ICS definitions(29)) and completed 3 day voiding diary demonstrating at least 1 episode of non-stress based urinary incontinence over the 72hr period (this may be urgency based incontinence or unaware incontinence).
* Patient is able to read and speak English

Exclusion criteria:

Based on Screening visit history:

* Participation in another drug or device study in the 60 days prior to the screening visit.
* Previous urologic surgery: Transurethral prostatectomy, bladder augmentation, sphincterotomy, bladder neck sling, artificial urinary sphincter, catheterizable channel, implantable electrostimulator/neuromodulator
* Current use of suprapubic catheter/foley catheter
* Unstable cardiac disease (uncontrolled hypertension, myocardial infarction, unstable angina, severe congestive heart failure (NYHA 3 or 4), ventricular arrhythmia (such as torsades de pointes), or stroke within the last 6 months)
* Clinically significant abnormal ECG
* The investigator believes the patient has an increased risk of QT prolongation (based on review of the screening ECG and patients concurrent medications)
* History of significant renal dysfunction within 1 year, or serum creatinine >150umol/L at screening visit (visit 1).
* History of significant liver disease within 1 year, or serum AST/ALT >2 times upper limit of normal, GGT >3 times upper limit of normal, total bilirubin >2 times upper limit of normal at screening visit (visit 1).
* History of pelvic radiation
* History of bladder cancer
* History of a concurrent malignancy or cancer (except noninvasive skin cancer) within the last 5 years. Subjects with a history of cancer are considered eligible if the subject has undergone potentially curative therapy and the subject has been considered disease free for at least 5 years (with the exception of basal cell or squamous cell carcinoma of the skin).
* Patient has a history of interstitial cystitis/pelvic pain syndrome
* Patient has a history of acute or chronic urinary retention within the last 3 months, and is currently not using intermittent catheters
* Patient has a history of a tachyarrhythmia
* Patient has a history of glaucoma
* Patient has a medical condition that may cause noncompliance with the study protocol
* In the opinion of the Investigator the patient has a history of significant stress urinary incontinence
* Patient has signs and symptoms of an active urinary tract infection (symptoms of dysuria, foul smelling urine, cloudy urine, increased spasticity, increased autonomic dysreflexia, self reported fever, increased incontinence, back/suprapubic pain).

  o Patient will submit urine for culture and sensitivity, undergo treatment, and will be eligible for rescreening after treatment.
* Female patient who is pregnant or breastfeeding, or plans to become pregnant.
* Male patient who is planning on fathering a child during the study or for 28 days after the last dose of study drug, or who is planning to donate sperm
* Patient refuses to provide written consent
* Patient will be unable or unwilling to complete the questionnaires and study visits
* In the opinion of the study investigator, it is not in the patient's best interest to be enrolled in this study.

Based on medication and allergy review

* The new addition of an anticholinergic medication, or a change to anticholinergic dose, within the last 30 days, (bladder specific anticholinergics include oxybutynin, tolterodine, fesoterodine, solifenacin, darifenacin, trospium, hyoscine, oxybutynin gel or patch, atropine, benzatropine). If previously used and discontinued, these medications must have been stopped for >2 weeks
* Newly added bladder active medication (or dose change) within the last 2 months (Tamsulosin, Silodosin, Terazosin, Baclofen, Diazepam, amitriptyline, Finasteride, Dutasteride, DDAVP/desmopressin)
* Use of flecainide, propafenone, donepezil, thioridazine, tramadol, aripiprazole, desipramine, imipramine, venlafaxine or digoxin
* Intravesical onabotulinum toxin use within the last 1 year
* Intravesical oxybutynin within the last 3 months
* Patient has a previous history of treatment with mirabegron
* Patient has a known allergy to mirabegron or a previous adverse reaction to a beta 3 agonist.

Based on physical exam

* Patient has a postvoid residual > 250mL at study enrollment after repeated tested (1 attempt to re-void to ensure complete emptying of the bladder) and is not using intermittent catheters
* Patient has a resting BP >180 mmHg systolic and/or >110 mmHg diastolic after 2 minutes of sitting quietly
* Patient has a resting heart rate >100bpm after 2 minutes of sitting quietly
* In the opinion of the study investigator, it is not in the patient's best interest to be enrolled in this study based on a clinically significant abnormality on physical exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blayne Welk, MD MSc, Principal Investigator — Western University
Locations (5):
- Canada (5):
  - Rehabiliation Center, Health Sciences Center, Winnipeg, Manitoba
  - Kingston General Hospital and Hotel Dieu Hospital (Queens University), Kingston, Ontario
  - Western University, London, Ontario
  - University of Ottawa, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mirabegron | Placebo
Started | 16 | 16
Completed | 15 | 14
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 14 | 15 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [43 to 58] | 56 [42 to 65] | 54 [42 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 8 | 9 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of participants with a Spinal cord injury (SCI), n [Count of Participants; unit: Participants] | 9 | 10 | 19
Number of participants with Mulitple sclerosis (MS), n [Count of Participants; unit: Participants] | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Bladder Capacity
Description: Urodynamic bladder capacity
Time Frame: 10 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 16 | 16
mL | 305 [234 to 376] | 369 [298 to 440]

2. Secondary Outcome: 3 Day Voiding Diary
Description: The 3 day voiding diary is a simple patient maintained record of fluid intake, voided volume and incontinence episodes. This will be used to assess number of episodes of urgency incontinence, urinary frequency, longest time between voids, functional capacity, and mean voided volume
Time Frame: 10 weeks
Reporting Status: Not Posted

3. Secondary Outcome: 24hr Urinary Pad Weights
Description: This will determine the amount of urinary incontinence that occurs over a 24hr period.
Time Frame: 10 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Quality of Life (Bladder Specific)
Description: The Short Form-Qualiveen is a urinary specific quality of life measure developed and studied specifically for neurogenic bladder patients; validity, reliability and responsiveness have been established.
Time Frame: 10 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Life (Incontinence)
Description: The I-QOL is an incontinence specific quality of life tool that has been shown to be a valid, reliable and responsive measurement among patients with neurogenic bladder dysfunction
Time Frame: 10 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Patient Reported Outcome Measure-NBSS
Description: The Neurogenic bladder symptom score (NBSS) is a symptom specific measure of urinary symptoms developed for patients with neurogenic bladder dysfunction with demonstrated validity and reliability. Minimum score is 0, maximum score is 74. Higher score is worse neurogenic bladder symptoms.
Time Frame: 10 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Patient Perception of Bladder Condition
Description: The patient perception of bladder condition is a commonly used measure in the assessment of oral medications for the treatment of overactive bladder symptoms
Time Frame: 10 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Adverse Events
Description: Adverse events will be monitored passively. They will be actively monitored for hypertension, tachycardia, and urinary retention.
Time Frame: 10 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Secondary Urodynamic Characteristics: Maximum Detrusor Pressure
Time Frame: 10 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Secondary Urodynamic Characteristics: Volume at Maximum Detrusor Pressure
Time Frame: 10 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Secondary Urodynamic Characteristics: Bladder Sensation
Time Frame: 10 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Secondary Urodynamic Characteristics: Bladder Compliance
Time Frame: 10 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Secondary Urodynamic Characteristics: Volume at First Detrusor Overactivity
Time Frame: 10 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 Weeks
Arm/Group | Mirabegron | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-09-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT02044510/Prot_SAP_000.pdf
  • Informed Consent Form (2014-09-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT02044510/ICF_001.pdf